CLINICAL TRIAL: NCT04759846
Title: 'An Open Label, Multicentre, Phase I Study to Evaluate the Impact of Moderate and Severe Hepatic Impairments on the Pharmacokinetics and Safety of Encorafenib in Combination With Binimetinib in Adult Patients With Unresectable or Metastatic BRAF V600-mutant Solid Tumors'.
Brief Title: Hepatic Impairment Study of Encorafenib in Combination With Binimetinib in BRAF Melanoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: no recruitment
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: W00090GE101
Record Dates: First submitted 2020-12-21; First posted 2021-02-18 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: BRAF V600 Mutation; Unresectable Melanoma; Metastatic Melanoma; Hepatic Impairment
MeSH Terms: conditions — Melanoma | interventions — encorafenib; binimetinib

STUDY DESIGN:
Intervention Model Description: Participants with hepatic impairment will be enrolled sequentially according to their severity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group with normal hepatic function (Experimental): Normal hepatic function
  Interventions: Drug: Encorafenib + Binimetinib
- Group with moderate hepatic impairment (Experimental): Moderate hepatic impairment (Child-Pugh Class B)
  Interventions: Drug: Encorafenib + Binimetinib
- Group with severe impairment (Experimental): Severe impairment (Child-Pugh Class C)
  Interventions: Drug: Encorafenib + Binimetinib

INTERVENTIONS:
Drug: Encorafenib + Binimetinib — The doses administered to patients with normal hepatic function will be the same as the recommended commercialised doses
  Other Names: Braftovi + Mektovi
  Arms: Group with normal hepatic function
Drug: Encorafenib + Binimetinib — A smaller dose than the dose approved for patients with normal hepatic function has been defined
  Other Names: Braftovi + Mektovi
  Arms: Group with moderate hepatic impairment
Drug: Encorafenib + Binimetinib — A smaller dose than the dose approved for patients with normal hepatic function has been defined
  Other Names: Braftovi + Mektovi
  Arms: Group with severe impairment

SUMMARY:
Encorafenib in combination with binimetinib have been approved in USA, Europe, Australia, Japan and Switzerland for the treatment of adult patients with unresectable or metastatic melanoma with BRAF V600 mutation.

The main objective of this study is to find a safe and effective dose of encorafenib in combination with binimetinib for patients who have BRAF-mutant metastatic or unresectable melanoma with hepatic dysfunction (i.e. moderate or severe impairment).

DETAILED DESCRIPTION:
This is an open label, multicentre, phase I study to evaluate the impact of moderate and severe hepatic impairment (HI) on the pharmacokinetics and safety of encorafenib in combination with binimetinib, in adult patients with unresectable or metastatic BRAF V600-mutant melanoma.

For each participant, the treatment period will be split in 2 phases:

* a HI assessment phase assessing the impact of hepatic impairment after a single dose (Day 1) and after repeated doses (Day 15).
* a post-HI assessment phase: after completing the HI assessment phase, participants may continue treatment in the post-HI assessment phase until disease progression or unacceptable toxicity.

Participants with hepatic impairment will be enrolled sequentially according to their severity. The study will start first in participants with normal hepatic function and moderate hepatic impairment respectively.

Participants will be assigned to one of the following 3 study groups:

* Group with normal hepatic function: 4 participants
* Group with moderate hepatic impairment (Child-Pugh Class B): 4 participants
* Group with severe impairment (Child-Pugh Class C): 4 participants

An Internal Review Committee (IRC) will review the safety and PK data of encorafenib in combination with binimetinib for group with normal hepatic function and group with moderate hepatic impairment and make a recommendation prior to start group with severe impairment enrolment. The Sponsor will determine whether it is safe and feasible to proceed with group with severe impairment.

Participants will receive treatment doses according to their assigned group.

ELIGIBILITY:
Inclusion Criteria

Participants must meet all of the following inclusion criteria to be eligible for enrolment into the study:

1. Signed written informed consent;
2. Male or female participant, aged ≥ 18 years;
3. Histologically/cytologically confirmed diagnosis of locally advanced, unresectable or metastatic solid tumors;
4. Presence of BRAF V600E or V600K mutation in tumour tissue prior to enrolment, as previously determined using a local test at any time prior to Screening - Only PCR and NGS-based local assays results will be acceptable;
5. Evidence of measurable or non-measurable lesions as detected by radiological or photographic methods according to guidelines based on Response Evaluation Criteria in solid tumors (RECIST) v. 1.1;
6. Unresectable locally advanced or metastatic solid tumor with no prior treatment or progression on or after prior systemic therapy; Note: Prior therapy with a BRAF inhibitor is permitted except in the regimen immediately prior to study entry. Progression during prior BRAF/MEK inhibitor treatment is not required;
7. Blood pressure (BP; after 5 minutes resting in the supine position) at screening within the following ranges: systolics, 90 to 150 mm Hg, diastolic, 50 to 100 mm Hg;
8. ECOG PS of 0 or 1;
9. Adequate bone marrow, organ function and laboratory parameters:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L,
   2. Haemoglobin (Hgb) ≥ 9 g/dL without transfusions,
   3. Platelets (PLT) ≥ 100 x 109/L without transfusions,
   4. International normalized ratio (INR) < 3 at screening or baseline (Day -1),
   5. Creatinine ≤ 1.5 mg/dL and calculated creatinine clearance (determined as per Cockcroft-Gault) ≥ 50 mL/min,
10. Hepatic function criteria:

    * Inclusion criteria for participant with normal hepatic function (group I) only :

      1. Total bilirubin ≤1.5 upper limit of normal (ULN) at screening and baseline (Day -1)
      2. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma- glutamyl transferase, and alkaline phosphatase ≤ 1.5ULN at screening and baseline (Day -1)
      3. Serum amylase <140 and lipase < 160ULN at screening and baseline (Day -1)
    * Inclusion Criteria for participants with Hepatic impairment according to Child-Pugh

    Classification System only:
    * Group II: Child-Pugh Class B or moderate hepatic impairment (7 to 9 points),
    * Group III: Child-Pugh Class C or severe hepatic impairment (10 to 15 points),
11. Able to take oral medications
12. Deemed by the Investigator to have the initiative and means to be compliant with the protocol (treatment and follow-up);
13. Female participant of childbearing potential must be tested negative for pregnancy at enrolment and during the study: Note: Negative serum beta-human chorionic gonadotropin (β-HCG) test (childbearing performed within 72 hours prior to first dose and consent to ongoing urine pregnancy testing during the course of the study and agreement to go on using it during the whole duration of the study and up to 1 month after last administration. Use of an effective method of contraception (hormonal contraception or intra-uterine device) assessed by the Investigator, for at least 2 months before the first study treatment administration, and agreement to go on using it in addition to condom during the whole duration of the study through 30 days after last study treatment administration.
14. Male participants with partners of childbearing potential must be either vasectomized or agree to use a condom in addition to having their partners use of an effective method of contraception. Note: For partner of male participant, contraception should be employed from the time of consent through 90 days after last study treatment administration.
15. Affiliated to a social security system, or is a beneficiary (if applicable in the national regulation)

Exclusion Criteria

Participants meeting any of the following criteria are not eligible for enrolment in the study:

1. A calculated Child-Pugh score that showed impairment for a reason other than liver dysfunction (e.g., cancer, cachexia);
2. History or symptoms of encephalopathy (Grade II or worse) within 4 weeks of Day -1 or subjetcs who were treated to control encephalopathy within 4 weeks of Day -1;
3. Clinical evidence of severe ascites (NCI-CTCAE grade 3 or 4);
4. History of surgical portosystemic shunt with complications (i.e., hepatic encephalopathy, heart failure). Trans jugular intrahepatic portosystemic shunt could have been allowed if not in use for ≥1 year;
5. Active bleeding during the last 28 days prior to dosing including variceal bleeding;
6. Anticoagulant therapy within 7 days prior to the first dose of study treatment (Day 1);
7. Any of the following:

   1. Nitrosourea or mitomycin-C within 6 weeks prior to start of study treatment,
   2. Other chemotherapy, radiation therapy that included > 30% of the bone, marrow reserve, or biological therapy (e.g., antibodies) within 4 weeks prior to start of study treatment,
   3. Continuous or intermittent small-molecule therapeutics or investigational agents within 5 half-lives of the agent or within 2 weeks prior to start of study treatment, whichever is the longest,
   4. Residual Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 side effects of any such therapy (residual Grade 2 alopecia is permitted),
8. Discontinuation of prior BRAF and/or MEK inhibitor treatment due to severe, intolerable toxicity including left ventricular dysfunction, pneumonitis/interstitial lung disease, or retinal vein occlusion, CK elevation and rhabdomyolysis, uveitis;
9. Symptomatic brain metastasis; Note: Participants previously treated or untreated for these conditions who are asymptomatic in the absence of corticosteroid and anti-epileptic therapy are allowed. Brain metastases must be stable for ≥ 4 weeks, with imaging (e.g., magnetic resonance imaging [MRI] or computed tomography [CT] demonstrating no current evidence of progressive brain metastases at screening);
10. Leptomeningeal disease;
11. Use, within 2 weeks prior to the first dose of the study treatment (Day 1)any herbal medications/supplements or any medications or foods that are moderate or strong inhibitors or inducers of CYP3A4/5;
12. Human immunodeficiency virus (HIV) infection;
13. Active viral hepatitis (HBV-HCV) within 1 month before the first dose of study treatment (Day 1);
14. Known history of acute or chronic pancreatitis;
15. Concurrent neuromuscular disorder that is associated with the potential of elevated creatine kinase (CK) (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy;
16. History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes);
17. Clinically significant cardiac disease including any of the following:

    1. Congestive heart failure requiring treatment (New York Heart Association Grade ≥ 2),
    2. Left ventricular ejection fraction (LVEF) < 50% as determined by MUGA or ECHO,
    3. Uncontrolled hypertension defined as persistent systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg despite current therapy,
    4. History or presence of clinically significant ventricular arrhythmias or atrial fibrillation,
    5. Clinically significant resting bradycardia,
    6. Unstable angina pectoris ≤ 3 months prior to the start of study treatment,
    7. Acute myocardial infarction ≤ 3 months prior to the start of study treatment,
    8. Mean triplicate QT interval corrected for heart rate using Fridericia's formula (QTcF) value >480 msec,
18. Impaired gastrointestinal function or disease which may significantly alter the absorption of study treatments (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhoea, malabsorption syndrome, small bowel resection);
19. History of chronic inflammatory bowel disease or Crohn's disease requiring medical intervention (immunomodulatory or immunosuppressive medications or surgery) ≤12 months prior to to starting study treatment the first dose of study treatment (Day 1);
20. Thromboembolic event (e.g. including transient ischemic attacks, cerebrovascular accidents, deep vein thrombosis or pulmonary emboli) except catheter-related venous thrombosis ≤ 12 weeks prior to starting study treatment (Day 1); Note: Participants with catheter-related thromboembolic events are allowed;
21. Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study treatment administration or that may interfere with the interpretation of study results and, in the judgement of the Investigator, would make the participant inappropriate for the study;
22. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until termination of gestation, confirmed by a positive β- hCG laboratory test (> 5 mIU/mL);
23. Known hypersensitivity or contraindication to any component of study treatment or their excipients;
24. Ongoing/active participation in another interventional clinical trial;
25. Has participated in another clinical trial with the administration of an investigational product within 4 weeks, or five times the half-life of the investigational product, whichever is longer, before the first dose of study treatment (Day 1);
26. Is a family member of the Investigator or any associate, colleague, and employee assisting in the conduct of the study (secretary, nurse, technician…).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Encorafenib Cmax | Day 1 and Day 15: 0-8 hours post-dose
  Maximum Observed Plasma Concentration of encorafenib expressed as total and unbound concentrations
Encorafenib AUClast | Day 1 and Day 15: 0-8 hours post-dose
  Area Under the Plasma Concentration versus Time Curve from Time 0 to Time of Last Quantifiable Concentration of encorafenib expressed as total and unbound concentrations
Encorafenib AUC(0-inf) | Day 1 and Day 15: 0-8 hours post-dose
  Area Under the Plasma Concentration versus Time Curve from Time 0 to Infinity of encorafenib expressed as total and unbound concentrations

SECONDARY OUTCOMES:
Tmax | Day 1 and Day 15: 0-8 hours post-dose
  Time to Reach Maximum Plasma Concentration of encorafenib and its metabolite (LHY746) and binimetinib and its active metabolite (AR00426032)
Cmin | Derived on Day1 and Day15
  Minimum Observed Plasma Concentration of encorafenib and its metabolite (LHY746) and binimetinib and its active metabolite (AR00426032) expressed as total and unbound concentrations
T1/2 | Day 1 and Day 15: 0-8 hours post-dose
  Terminal Phase Plasma Half-life of encorafenib and binimetinib and their metabolite
CL/F | Day 1 and Day 15: 0-8 hours post-dose
  Apparent Total Body Clearance of encorafenib and binimetinib and their metabolites as total and unbound concentrations
Vz/F | Day 1 and Day 15: 0-8 hours post-dose
  Apparent Volume of Distribution at Terminal Phase of encorafenib and binimetinib and their metabolites as total and unbound concentrations
MRCmax | Derived on Day1 and Day15
  Metabolic Ratio of Cmax of LHY746 to Cmax of encorafenib, Metabolic Ratio of Cmax of AR00426032 to Cmax of binimetinib Corrected for Molecular Weights
MRAUC | Derived on Day1 and Day15
  Metabolic Ratio of AUC of LHY746 to AUC of encorafenib, Metabolic Ratio of AUC of AR00426032 to AUC of binimetinib Corrected for Molecular Weights

CONTACTS AND LOCATIONS:
Overall Officials: Petr Arenberger, Principal Investigator — Fakultni Nemocnice Kralovske Vinohrady, Czech Republic
Locations (7):
- Czechia (2):
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni Nemocnice Kralovske Vinohrady, Prague
- Italy (2):
  - Irccs Irst, Meldola
  - Azienda Ospedaliero, Siena
- Spain (3):
  - all D'Hebron Insitute of Oncology, Barcelona
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital General de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No